CLINICAL TRIAL: NCT02823834
Title: Post Market Clinical Follow-up Study Protocol for PROFEMUR® Gladiator Plasma Femoral Stems and PROCOTYL® L Beaded Acetabular Components
Brief Title: PMCF Study Protocol for PROFEMUR® Gladiator Plasma Femoral Stems and PROCOTYL® L Beaded Acetabular Components
Status: Active, not recruiting | Type: Observational
Sponsor: MicroPort Orthopedics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-LJH-002H
Record Dates: First submitted 2016-07-01; First posted 2016-07-06 (Estimated); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Joint Disease
Keywords: osteoarthritis; avascular necrosis; ankylosis; protrusio acetabuli; painful hip dysplasia; rheumatoid arthritis; correction of functional deformity
MeSH Terms: conditions — Joint Diseases; Osteoarthritis; Osteonecrosis; Ankylosis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PROFEMUR® Gladiator Plasma Femoral Stems: Single study group either previously implanted with the following combination of components: PROFEMUR® Gladiator Plasma Femoral Stems, PROCOTYL® L Beaded Acetabular Shells, Polyethylene or Ceramic Liners, and Metal or Ceramic Femoral Heads.
  Interventions: Device: PROFEMUR® Gladiator Plasma Femoral Stems

INTERVENTIONS:
Device: PROFEMUR® Gladiator Plasma Femoral Stems — THA using PROFEMUR® Gladiator Plasma stems and PROCOTYL® L Beaded Acetabular Components
  Other Names: Primary hip replacement device

SUMMARY:
MicroPort Orthopedics (MPO) is conducting this post market clinical follow-up (PMCF) study to evaluate the safety and efficacy of its total hip arthroplasty (THA) components marketed in the European Union (EU). These types of studies are required by regulatory authorities for all THA devices that do not have medium to long-term clinical evidence available at the time of gaining approval to market in the EU. This study has been designed in accordance with the medial device directives (MEDDEV) 2.12/2 rev 2.

ELIGIBILITY:
Inclusion Criteria:

* Has undergone primary THA for any of the following:
* Non-inflammatory degenerative joint disease such as osteoarthritis, avascular necrosis, ankylosis, protrusio acetabuli, or painful hip dysplasia;
* Inflammatory degenerative joint disease such as rheumatoid arthritis; or
* Correction of functional deformity
* Subject is implanted with the specified combination of components
* Subject is willing and able to complete required study visits or assessments

Previously implanted bilateral subjects can have both THAs enrolled in the study provided:

* the specified combination of components were implanted in both
* all other aspects of the Inclusion/Exclusion Criteria are satisfied
* enrollment does not exceed the subject count specified in the Clinical Trial Agreement
* the subject agrees to a second Informed Consent document specific to the second THA.

Exclusion Criteria:

* Subjects implanted with a metal-on-metal articulation
* Subjects implanted with non-MPO or non-Wright Medical Technology components (femoral heads, acetabular shells, acetabular liners) at the time of their primary THA in the enrolled THA
* Subjects skeletally immature (less than 21 years of age) at time of primary THA surgery
* Subjects currently enrolled in another clinical study which could affect the endpoints of this protocol
* Subjects unwilling to sign the Informed Consent document
* Subjects with substance abuse issues
* Subjects who are incarcerated or having pending incarceration

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been previously implanted with a PROFEMUR® Gladiator Plasma Femoral Stem and PROCOTYL® L Beaded Acetabular Component
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Component Survivorship | 10 years post-operative
  The primary objective of this study is to estimate survivorship analysis of all components at specified intervals out to 10 years follow-up.

SECONDARY OUTCOMES:
Patient functional outcomes (hip specific) | 2-5 years, 5-7 years and 10 years postoperatively beginning with first available visit
  To characterize total functional scores, as assessed by Oxford Hip Scores
Patient functional outcomes (quality of life) | 2-5 years, 5-7 years and 10 years postoperatively beginning with first available visit
  To characterize total functional scores, as assessed by EQ-5D-3L scores

CONTACTS AND LOCATIONS:
Overall Officials: Jose Pimienta, Principal Investigator — Elbe Kliniken Buxtehude
Locations (1):
- Elbe Kliniken Buxtehude, Buxtehude, Germany

IPD SHARING:
Plan to Share IPD: No